CLINICAL TRIAL: NCT01091792
Title: DMS 0947 Exploratory Study of the Modulation of the Immune System by Vascular Endothelial Growth Factor (VEGF) Blockade in Patients With Glioblastoma Multiforme (GBM)
Brief Title: Exploratory Study of the Modulation of the Immune System by VEGF Blockade in Patients With Glioblastoma Multiforme (GBM)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Lionel.D.Lewis, MD, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D0947
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM; Grade IV; glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): Bevacizumab + temozolomide + radiotherapy followed by adjuvant bevacizumab + temozolomide
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab every 2 weeks 10mg/kg beginning 2 weeks after start of Radiation Therapy
  Other Names: Avastin

SUMMARY:
Blood samples will be obtained from newly diagnosed GBM patients treated with combined radiotherapy (RT), temozolomide (TMZ) and bevacizumab (BEV) at specific time points. The primary outcome is the shift in T reg cell fraction a defined by determining the proportion of CD4 cells that are CD4+ CD25.

DETAILED DESCRIPTION:
Glioblastoma multiforme (GBM) is the most frequent malignant brain tumor and it remains a lethal disease. Approximately 4 weeks post surgery for tumor resection, patients will proceed to standard of care treatment which currently consists of temozolomide (TMZ) with concurrent radiation therapy (RT) for 6 weeks. This study will add bevacizumab (BEV) to the standard of care regimen in newly diagnosed patients. The Bevacizumab will be added 2 weeks post start of RT/TMZ. Administration of bevacizumab will continue concurrently with TMZ every 2 weeks for 12 months. Blood samples will be obtained from these patients at 3 different time points during this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven GBM
* Karnofsky status equal to or greater than 60%

Exclusion Criteria:

* Inadequately controlled hypertension
* Prior history of hypertension crisis or hypertensive encephalopathy
* History of stroke or transient ischemic attach within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-03; Primary Completion 2015-04-02 (Actual); Study Completion 2015-04-02 (Actual)

PRIMARY OUTCOMES:
Changes in the peripheral blood T-reg profile between pretreatment and 4 weeks after completion of treatment with the addition of bevacizumab to RT and TMZ in patients with glioblastoma | 1 year

SECONDARY OUTCOMES:
Immunologic shift in the phenotypic T cell, B cell, NK cell and DC repertoire induced by RT-TMZ-BEV comparing pretreatment and 4 weeks after completion of treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Camilo E Fadul, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hithcock Medcial Center, Lebanon, New Hampshire, United States